CLINICAL TRIAL: NCT01710098
Title: Effectiveness and Safety as Well as Adherence of the "S3 Guidelines for the Treatment of Prostate Cancer" in the Treatment of Patients of Patients With Firmagon®
Brief Title: Treatment of Prostate Cancer With Firmagon®
Status: Completed | Type: Observational
Sponsor: United Clinic Management GmbH (Industry)
Responsible Party: Principal Investigator, Karin Buchsteiner, Head of Study Group, United Clinic Management GmbH
Other Study IDs: UCM12-01
Record Dates: First submitted 2012-10-10; First posted 2012-10-18 (Estimated); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Prostate Cancer
Keywords: testosterone; S3-Adherence; Quality of Life
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Degarelix: adult male patients with advanced hormone dependent prostate cancer who receive 240 mg as a start dose and then monthly 80mg Firmagon® for one year
  Interventions: Drug: Degarelix

INTERVENTIONS:
Drug: Degarelix — subcutaneous injection
  Other Names: Firmagon®

SUMMARY:
How are testosterone levels of patients with prostate cancer under treatment with Firmagon® changing.

Former studies showed a quick fall of testosterone levels after start of therapy with Firmagon® and a quick recovery when therapy is stopped. The investigators want to prove this in a normal outpatient urologist setting. Furthermore data is collected to prove the adherence to the German S3-Guideline for the treatment of prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* advanced hormone-dependent prostate cancer with no other previous hormone therapy for whom - irrespectively of this NIS -the use of Firmagon® is intended

Exclusion Criteria:

* contraindication for Degarelix

Ages: 18 Years to 95 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult male patients of outpatient urological medical practice
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-06; Primary Completion 2014-06 (Actual); Study Completion 2015-09-24 (Actual)

PRIMARY OUTCOMES:
PSA-/Testosterone Level | 12 months

SECONDARY OUTCOMES:
S3 Guideline | 12 months
  Percentage of patients who have been treated in accordance with the grade A recommendations of the S3 guideline for treatment of prostate cancer
Anxiety | 12 Months
  Anxiety score

CONTACTS AND LOCATIONS:
Overall Officials: Leopold Durner, MD, Principal Investigator — UCM GmbH
Locations (1):
- UCM GmbH, Planegg, Bavaria, Germany

REFERENCES:
- [Background] Thompson IM, Zeidman EJ, Rodriguez FR. Sudden death due to disease flare with luteinizing hormone-releasing hormone agonist therapy for carcinoma of the prostate. J Urol. 1990 Dec;144(6):1479-80. doi: 10.1016/s0022-5347(17)39774-4. PMID 2122011
- [Background] Klotz L, Boccon-Gibod L, Shore ND, Andreou C, Persson BE, Cantor P, Jensen JK, Olesen TK, Schroder FH. The efficacy and safety of degarelix: a 12-month, comparative, randomized, open-label, parallel-group phase III study in patients with prostate cancer. BJU Int. 2008 Dec;102(11):1531-8. doi: 10.1111/j.1464-410X.2008.08183.x. PMID 19035858
- [Background] Morote J, Orsola A, Planas J, Trilla E, Raventos CX, Cecchini L, Catalan R. Redefining clinically significant castration levels in patients with prostate cancer receiving continuous androgen deprivation therapy. J Urol. 2007 Oct;178(4 Pt 1):1290-5. doi: 10.1016/j.juro.2007.05.129. Epub 2007 Aug 14. PMID 17698136
- [Background] Perachino M, Cavalli V, Bravi F. Testosterone levels in patients with metastatic prostate cancer treated with luteinizing hormone-releasing hormone therapy: prognostic significance? BJU Int. 2010 Mar;105(5):648-51. doi: 10.1111/j.1464-410X.2009.08814.x. Epub 2009 Aug 28. PMID 19747358
- [Background] Mariani S, Salvatori L, Basciani S, Arizzi M, Franco G, Petrangeli E, Spera G, Gnessi L. Expression and cellular localization of follicle-stimulating hormone receptor in normal human prostate, benign prostatic hyperplasia and prostate cancer. J Urol. 2006 Jun;175(6):2072-7; discussion 2077. doi: 10.1016/S0022-5347(06)00273-4. PMID 16697805
- [Background] Radu A, Pichon C, Camparo P, Antoine M, Allory Y, Couvelard A, Fromont G, Hai MT, Ghinea N. Expression of follicle-stimulating hormone receptor in tumor blood vessels. N Engl J Med. 2010 Oct 21;363(17):1621-30. doi: 10.1056/NEJMoa1001283. PMID 20961245
- [Background] Heidenreich A., Epplen R., Thüer D., Van Erps T., D.P., EURO Prostate Center. EAU guideline on advanced prostate cancer: Compliance among urologists conderning androgen deprivation therapy